CLINICAL TRIAL: NCT03914235
Title: Efficacy of Tumescent Local Anesthesia in the Surgical Management of Tenosynovitis.
Brief Title: Anesthesia Tumescent for Surgical Management of Tenosynovitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, Investigador de tiempo completo, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2018-1301-021
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Tenosynovitis
Keywords: Tumescent anesthesia; tenosynovitis; Visual Analog Scale; Tourniquets; Epinephrine
MeSH Terms: conditions — Tenosynovitis | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tumescent anesthesia (Experimental): A tumescent solution was prepared; consisting of 40 cc of 0.9% Saline Solution, 10 cc of 2% Lidocaine, 0.4 cc of Epinephrine (1: 1000) and 4 cc of 7.5% Sodium Bicarbonate. This solution was applied in the incision sites according to the diagnosis and the proposed procedure. In case of trigger finger, 3 cc was applied subcutaneously in the proximal palmar crease of the affected finger; for Quervain syndrome, 5 to 6 cc of tumescent solution was injected along the first extensor compartment at the radial styloid level; and in the case of Carpal Tunnel Syndrome, 10 cc of tumescent solution was infiltrated on the flexor retinaculum in the subcutaneous tissue and from 7 to 10 cc below it. Subsequently, 20 minutes were waited for the epinephrine to cause vasoconstriction, and the asepsis of the limb was continued , sterile fields were placed, the incision site was corroborated and the surgical procedure proposed for each pathology was started.
  Interventions: Combination Product: Tumescent Anesthesia; Procedure: Open release of the tendon
- Local anesthesia with tourniquet. (Active Comparator): Lidocaine 1% was applied to the incision sites according to the diagnosis and the proposed procedure. In case of trigger finger, 3 cc was applied subcutaneously in the proximal palmar crease of the affected finger; for Quervain syndrome, 5 to 6 cc were injected along the first extensor compartment at the radial styloid level; and in the case of Carpal Tunnel Syndrome, 10 cc was infiltrated on the flexor retinaculum in the subcutaneous tissue and from 7 to 10 cc below it. Afterwards, a pneumatic tourniquet was placed at the level of the forearm at 250 mmHg after exsanguination with a bandage from Esmarch. The asepsis of the limb was continued, sterile fields were placed, the incision site was corroborated and the surgical procedure proposed for each pathology was started.
  At the end of the surgical procedure, it was closed by planes, a soft bandage was placed, the tourniquet was removed and the patient was taken to recovery.
  Interventions: Drug: Lidocaine; Device: Pneumatic tourniquet; Procedure: Open release of the tendon

INTERVENTIONS:
Combination Product: Tumescent Anesthesia — A tumescent solution is prepared with 2% lidocaine (10ml), 1:1000 epinephrine (0.4ml) and 7.5% sodium bicarbonate (4ml) dissolved in 0.9% saline solution (40ml) and applied from 3 to 20ml (depending on the pathology to be repaired) at the incision site.
  Arms: Tumescent anesthesia
Drug: Lidocaine — Apply 3 to 20 ml at the incision site, depending on the pathology to be repaired(carpal tunnel syndrome, trigger finger or Quervain syndrome).
  Other Names: Lidocaine 1%
  Arms: Local anesthesia with tourniquet.
Device: Pneumatic tourniquet — Level of the forearm at 250 mmHg, after exsanguination with Esmarch bandage.
  Arms: Local anesthesia with tourniquet.
Procedure: Open release of the tendon — Standard surgical procedure for carpal tunnel syndrome, trigger finger and Quervain syndrome.

SUMMARY:
The aim of this study is to evaluate the effectiveness of the tumescent anesthesia technique in the surgical management of hand tenosynovitis. For this, an open clinical trial was conducted, which included patients with hand tenosynovitis (carpal tunnel syndrome, trigger finger and Quervain syndrome), which were randomly assigned to a group. The control group was released pulleys and ligaments with local anesthetic technique and hemostasis with pneumatic tourniquet; While the study group was released from the pulleys and ligaments with tumescent anesthesia. The study variables were: anesthesia time, trans-surgical bleeding, pain, total procedure time and tissue reperfusion time.

DETAILED DESCRIPTION:
Introduction: The WALANT technique (Wide Awake Local Anesthesia No-Torniquet) proposes the use of local anesthesia, epinephrine and tourniquet in the areas of the hand to be repaired, making costs and time and comfort more efficient.

Objective: Evaluation of the effectiveness of the WALANT technique versus regional anesthesia with tourniquet in pain control, surgical management of stenosing tenosynovitis.

Material and methods: Open clinical trial including patients with the trigger finger, tunnel syndrome in the operating room, candidates for surgery, and excluding previous surgeries at the site of the injury, hemodynamic instability, peripheral vascular diseases, smoking, anxiety, or psychiatric diseases. The anesthetic method was applied to the incision sites according to the diagnosis and the proposed procedure. At the end of the test, tumescent solution and control, 1% lidocaine plus pneumatic tourniquet on the forearm at 250mmHg. The main variables were: type of anesthesia and pain during the procedure. Descriptive and inferential statistics were applied (xi2, t-student or Mann-Whitney U).

ELIGIBILITY:
Inclusion Criteria:

* Right holders of the Mexican Social Security Institute
* Over 18 years
* Trigger Finger Diagnosis
* Diagnosis of Carpal Tunnel Syndrome
* Diagnosis of Quervain Syndrome
* Acceptance and signature of informed consent

Exclusion Criteria:

* Necessity for concomitant surgery
* Previous surgeries on the injured site
* Hemodynamic instability
* History of peripheral vascular diseases
* Do not wish to participate in the study
* Hypersensitivity to medication
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Procedure pain: Visual Analog Scale | immediate post surgery
  Evaluated by Visual Analog Scale, A subjective psychometric response scale used to measure distinct behavioral or physiological phenomena based on linear numerical gradient, with values from 0 to 10. In the value 0 the absence or less intensity is located and in 10 the greater intensity of pain.

SECONDARY OUTCOMES:
Bleeding | immediate post surgery
  Bleeding estimated in consensus between anesthesiologist and surgeon, based on the gauze used during surgery
Anesthesia application time | at the beginning of the application of anesthesia
  The interval of time in minutes that is required to apply the anesthetic method chosen in the area to be used

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes Orozco, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No